CLINICAL TRIAL: NCT02377284
Title: Engaging Food Service Workers in the Prevention of Food Allergy-related Adverse Events
Brief Title: Prevention and Management of Food Allergies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Carolyn Cannuscio, Assistant Professor of Family Medicine and Community Health, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 818836
Record Dates: First submitted 2015-02-06; First posted 2015-03-03 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Empathy; Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Moire Topography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (personalized chef card) (Experimental): Restaurant employees received a personalized chef card, which included written information about a patron's food allergies and a photograph of the patron.
  Interventions: Other: Photograph
- Control (depersonalized chef card) (No Intervention): Restaurant employees received a depersonalized chef card, which included written information about a patron's food allergies, without a photograph of a patron.

INTERVENTIONS:
Other: Photograph — Add a photograph to a chef card.
  Arms: Intervention (personalized chef card)

SUMMARY:
This pilot study will test the use of visual cues to engage food service workers in protecting patrons with food allergies. Food service workers from Philadelphia quick-service restaurants were recruited to participate in a survey of attitudes that includes an embedded randomized experiment testing an experimental cue (photograph of an allergic child) to increase workers' engagement and empathy.

DETAILED DESCRIPTION:
Aim: Investigators pilot-tested a novel strategy to engage food service workers, by using a visual cue to increase the workers empathy for and desire to protect the patrons health and safety.

Why intervene with food service workers? Both food allergies and allergenic foods are common, as is eating, making accidental ingestion of allergenic foods almost inevitable. Risks may be particularly pronounced in out-of-home contexts (restaurants, school cafeterias, etc.), where the food allergic person must rely on service workers to assure their safety. Therefore, food service workers are important partners in the prevention of adverse events.

Design: Within the context of a survey of food service workers, investigators embedded a randomized experiment. In this experiment, investigators randomly assigned survey participants to one of two conditions: a Personalized vs. Depersonalized Chef Card. Depersonalized Chef Cards included simple written instructions regarding the patron's specific food allergies, including explicit guidance regarding foods to be avoided and information regarding the seriousness of the allergy. Personalized Chef Cards included identical written instructions and information, as well as a photograph of a patron with food allergies.

Hypothesis: Service workers exposed to the Personalized (compared to Depersonalized) Chef Cards will demonstrate greater empathy, sympathy, willingness to help, and vigilance regarding food allergies and their management.

ELIGIBILITY:
Inclusion Criteria:

* Employed at a quick-service restaurant
* Speaks English

Exclusion Criteria:

* Work at a table-only establishment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Mean knowledge and attitude scores reported by participants in both study groups | Investigators measured primary outcomes on Day 1 for each participant.
  Mean scores (on a scale from 0-100, assessed using a survey) for knowledge and attitudes regarding food allergic patrons among both the intervention and control groups.

SECONDARY OUTCOMES:
Mean empathy and desire to learn scores reported by participants in both study groups | Investigators measured secondary outcomes on Day 1 for each participant.
  Mean scores (on a scale from 0-100, assessed using a survey) for willingness to assist patrons with food allergies and desire to learn more about food allergies among both the intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn C Cannuscio, ScD, Principal Investigator — University of Pennsylvania

REFERENCES:
- [Result] Dupuis R, Meisel Z, Grande D, Strupp E, Kounaves S, Graves A, Frasso R, Cannuscio CC. Food allergy management among restaurant workers in a large U.S. city. Food control 63:147-57, 2016.